CLINICAL TRIAL: NCT04134247
Title: Study of PD-1 Monoclonal Antibody in Combination With Chemotherapy in Patients With Relapsed or Refractory Non-Hodgkin Lymphoma
Brief Title: Study of PD-1 Monoclonal Antibody in Combination With Chemotherapy in Patients With RR NHL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Xin, Director of Department of Hematology, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShandongPH006
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Relapsed/Refractory Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 combined with chemotherapy (Experimental): 21 days every cycle, assessment after 3-cycle
  Interventions: Drug: PD-1 combined with chemotherapy
- chemotherapy (Active Comparator): 21 days every cycle, assessment after 3-cycle
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Drug: PD-1 combined with chemotherapy — PD-1 200 mg，d1; Rituximab 375mg/m2，d0（ the same as the chemotherapy group）
  The chemotherapy chooses one of the following:
  GDP：Gemcitabine 800-1000mg/m2, d1、8; Cisplatin 25mg/m2, d1-3; Dexamethasone 40mg, d1-4; GemOx：Gemcitabine 800-1000mg/m2, d1、8; Oxaliplatin 130mg/m2，d1; DA-EPOCH：Epirubicin 15mg／m２ ,d1-4; Etoposide 50mg／m２ ,d1-4; Vincristine 0.4mg/ ｍ２ ，d1-4; Cyclophosphamide 750mg/ ｍ２ , d５; Prednisone 60mg/m２/d, d1-5; ICE: Ifosfamide 1g/m２，d1-4; Cisplatin 25mg/m２, d1-4; Etoposide 60 mg／m２，d1-4; DICE: Ifosfamide 1 g／m２，dl-d4; Cisplatin 25mg/m２, d1-4; Etoposide 60 mg／m２，d1-4; Dexamethasone 10-20mg，d1-4; High dose MTX（Central recurrence）：MTX 3.5g／ｍ２,ｄ1; Hyper CVAD（B）：MTX 1g／ｍ２, d1; Cytarabine 2-3g／ｍ２, q12h, d2-3
  Other Names: PD-1 combined with chemotherapy group
  Arms: PD-1 combined with chemotherapy
Drug: chemotherapy — Rituximab 375mg/m2，d0（ Except for patients who relapsed within12 months after the last application of rituximab）
  The chemotherapy chooses one of the following:
  GDP：Gemcitabine 800-1000mg/m2, d1、8; Cisplatin 25mg/m2, d1-3; Dexamethasone 40mg, d1-4; GemOx：Gemcitabine 800-1000mg/m2, d1、8; Oxaliplatin 130mg/m2，d1; DA-EPOCH：Epirubicin 15mg／m２ ,d1-4; Etoposide 50mg／m２ ,d1-4; Vincristine 0.4mg/ ｍ２ ，d1-4; Cyclophosphamide 750mg/ ｍ２ , d５; Prednisone 60mg/m２/d, d1-5; ICE: Ifosfamide 1g/m２，d1-4; Cisplatin 25mg/m２, d1-4; Etoposide 60 mg／m２，d1-4; DICE: Ifosfamide 1 g／m２，dl-d4; Cisplatin 25mg/m２, d1-4; Etoposide 60 mg／m２，d1-4; Dexamethasone 10-20mg，d1-4; High dose MTX（Central recurrence）：MTX 3.5g／ｍ２,ｄ1; Hyper CVAD（B）：MTX 1g／ｍ２, d1; Cytarabine 2-3g／ｍ２, q12h, d2-3
  Other Names: chemotherapy group
  Arms: chemotherapy

SUMMARY:
Lymphoma is one of the fastest growing malignancies in the world, with an annual incidence rate of about 4%. Non-Hodgkin's lymphoma (NHL) is highly heterogeneous and can be broadly divided into two major categories, B-cell lymphoma and T/NK cell lymphoma. It is composed of diseases of different pathological types and malignant degrees, and the prognosis is not the same.The anti-PD-1 antibody may benefit patients with relapsed or refractory Hodgkin's lymphoma. At the same time, in non-Hodgkin's lymphoma, PD1 antibodies also show promising therapeutic prospects. We propose this research program, based on the previous research at home and abroad, to further clarify the role of PD-1 monoclonal antibody combined with chemotherapy in the treatment of relapsed and refractory NHL patients, evaluate its clinical efficacy and safety, and explore The best treatment strategy for patients with relapsed and refractory NHL in China.

DETAILED DESCRIPTION:
Lymphoma is one of the fastest growing malignancies in the world, with an annual incidence rate of about 4%. In recent years, the incidence of malignant lymphoma in China has increased rapidly. It has risen to the ninth place among the top ten high-incidence tumors in men, and the female has risen to the eleventh place. In 2011, the incidence of lymphoma in the country has reached 6.43/100,000.

According to the characteristics of clinicopathology, lymphoma is divided into two categories: Hodgkin's lymphoma (HL) and non-Hodgkin's lymphoma (NHL). HL is a single disease, relatively rare, but the prognosis is good, and patients with limited period have no progress for 5 years. The survival rate was 85-95%, and the 5-year progression-free survival rate of advanced patients was 30-85%. NHL is highly heterogeneous and can be broadly divided into two major categories, B-cell lymphoma and T/NK cell lymphoma. It is composed of diseases of different pathological types and malignant degrees, and the prognosis is not the same.

In recent years, immunological checkpoint inhibitors have been the focus of research in the field of malignant tumor treatment. In clinical trials, PD-1/PD-L1 was found to be abnormally expressed in various lymphomas, including T-cell lymphoma, mediastinal large B-cell lymphoma, classical Hodgkin's lymphoma (CHL), and large variability. Cell lymphoma. Previous studies have evaluated the effects of antibody-based drugs against PD-1 (such as navobizumab and pabuleizumab) in patients with relapsed or refractory classic Hodgkin's lymphoma, and A higher response rate is shown and the security feature is acceptable. The domestic ORIENT-1 study showed that ididilimumab was highly active in patients with relapsed or refractory classic Hodgkin's lymphoma in China, and 80% (74/92) patients had an objective response. No patients died during the study. Of the 96 patients treated, 89 (93%) had treatment-related adverse events, including 17 (18%) patients with grade 3 or 4 treatment-related adverse events, and 11 patients (11%) experienced severe Adverse events, but no unexpected or off-target safety signals were found. Therefore, PD1 antibodies may benefit patients with relapsed or refractory Hodgkin's lymphoma.

At the same time, in non-Hodgkin's lymphoma, PD1 antibodies also show promising therapeutic prospects. Clinical studies at home and abroad have shown that PD-1 inhibitors are effective in relapsed or refractory extranodal NKT lymphoma. The results of the Idiliumab ORIENT-4 test showed that 1 year OS 82.1%, ORR 67.9%, DCR 85.7%, and PD-1 inhibitor combined with citabin to treat relapsed or refractory extranodal NKT is underway; PD-1 inhibitor monotherapy for relapsed or refractory PTCL is generally effective (ORR 33%, 4 of them CR); PD-1 inhibitor monotherapy is effective in treating relapsed or refractory mycosis/Sezary syndrome (ORR) 37.5%) has been recommended by the NCCN guidelines; trials in combination with IFN γ-1b are underway. PD-1 inhibitor monotherapy for relapsed or refractory PMBCL or PCNSL is effective, and PD-1 inhibitors have been recommended by the NCCN guidelines for the former treatment.

Therefore, we propose this research program, based on the previous research at home and abroad, to further clarify the role of PD-1 monoclonal antibody combined with chemotherapy in the treatment of relapsed and refractory NHL patients, evaluate its clinical efficacy and safety, and explore The best treatment strategy for patients with relapsed and refractory NHL in China.

ELIGIBILITY:
Inclusion Criteria:

1. Non-Hodgkin's lymphoma (NHL) confirmed by histopathology, preferably in the detection of tumor tissue PD-L1 expression.
2. A recurrent or refractory disease defined as: 1) recurrence of disease after complete remission (CR); or 2) partial remission (PR), disease stabilization (SD), or disease Progress (PD) when the treatment is completed prior to enrollment in the study.
3. Age≥18 years old, both men and women.
4. The ECOG score is 0-2.
5. There is at least one evaluable lesion (maximum diameter>15mm or shortest diameter>10mm). Preferably, PET-CT shows high metabolism of FDG.
6. Have received appropriate first-line and more-line treatment of the corresponding NHL.
7. Liver and kidney function: blood bilirubin≤35μmol/L, AST or ALT is less than 2 times the upper limit of normal value, serum creatinine≤150μmol/L.
8. The thyroid function is normal.
9. Women of childbearing age are required to undergo a pregnancy test before receiving treatment and must agree to take effective contraception during treatment.
10. Subjects must sign an informed consent form.

Exclusion Criteria:

1. Age<18 years old；
2. Received ASCT within 90 days prior to the first use of the study drug;
3. Severe allergies, or patients known to be allergic or intolerant of the drug components of the chemotherapy regimen;
4. Active, unrecognized or suspected autoimmune disease, or a history of autoimmune disease within 2 years;
5. Previously exposed to any antibody against PD-1, PD-L1 or cytotoxic T lymphocyte-associated antigen 4
6. Exposure to any study drug within 4 weeks prior to the first use of the study drug
7. Expose to the last radiotherapy or anti-tumor therapy (chemotherapy, targeted therapy, immunotherapy or arterial embolization) within 3 weeks prior to the first use of the study drug.
8. Have a history of oncology and have received any treatment for this tumor in the past 3 years;
9. Patients during pregnancy and lactation;
10. Accompanied by severe heart disease, including acute myocardial infarction within 6 months, or in accordance with New York Heart Association cardiac function III or IV;
11. A serological test for HIV or active hepatitis C virus is known to be positive;
12. Hepatitis B virus carriers or hepatitis B virus DNA positive untreated patients are known;
13. TB patients active period
14. Other circumstances that the investigator believes are not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 2 years
  Percentage of patients with complete remission （CR）or partial remission （PR）

SECONDARY OUTCOMES:
Progression free survival（PFS） | 2 years
  Time from enrollment to tumor progression or death
overall survival（OS） | 2 years
  Time from enrollment to death

CONTACTS AND LOCATIONS:
Overall Officials: Wang Xin, MD,PhD, Principal Investigator — Shandong Provincial Hospital
Locations (1):
- Department of Hematology, Shandong Provincial Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No